CLINICAL TRIAL: NCT02226471
Title: Serum CTRP3 and RBP4 Levels in Obesity and Hypertension
Status: Completed | Type: Observational
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Deng Wu Quan, Chongqing southwest hospital, Third Military Medical University
Other Study IDs: SW1000
Record Dates: First submitted 2014-08-24; First posted 2014-08-27 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Obesity; Hypertension
MeSH Terms: conditions — Obesity; Hypertension

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- NW-NBP group: normal weight and blood pressure subjects
- NW-HTN group: Normal weight with hypertension subjects
- OB-NBP group: obese-normal blood pressure subjects
- OB-HTN group: Obese-hypertension subjects

SUMMARY:
Insulin resistance is closely correlated with obesity and cardiovascular disease. Adipokines may play important roles in the pathogenesis of obesity, which are a link between obesity and obesity-related disorders.C1q/TNF-related protein-3 (CTRP3) and retinol-binding protein 4 (RBP4) are novel adipokine that modulates the action of insulin in various diseases. This study addressed the relationship between CTRP3, RBP4 and IR in newly diagnosed obesity and essential hypertension.

DETAILED DESCRIPTION:
Serum CTRP3 and RBP4, anthropometric and metabolic parameters were determined in 480 newly diagnosed obesity and essential hypertensive patients not taking anti-obese and antihypertensive medications and 66 normal weight (NW) and normotensive subjects. All subjects were divided into two groups depending on body mass index (BMI), including NW group and obesity group, and then four subgroups were divided according to obesity and hypertension, including NW-normal blood pressure subgroup (NW-NBP), NW-hypertension subgroup (NW-HTN), obese-normal blood pressure subgroup (OB-NBP), obese-hypertension subgroup (OB-HTN).

ELIGIBILITY:
Inclusion Criteria:

1. Hypertension not taking antihypertensive medications
2. Obesity not taking anti-obese or lipid-lowering medications

Exclusion Criteria:

1. Heart failure;
2. pregnant or lactating
3. diabetes
4. thyroid disease
5. fractures
6. osteoporosis
7. tumors;

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We consecutively selected 2100 Chinese subjects from the general population who had undergone medical check-ups at the Southwest Hospital Medical Center at the Third Military Medical University
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2012-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
CTRP3 and RBP4 levels were measured in obesity and hypertension | 1 year
  531 subjects were required to fast overnight before the physical examination.Blood pressure was measured three times, each 2 min apart on the upper arm using a mercury sphygmomanometer in a seated, resting position after 10 minutes of rest; the mean of the three measurements was used for the statistical analysis.Weight, height and hip and waist circumference (WC), were measured. BMI was calculated as body weight in kilograms divided by the square of height (m2). WHR was calculated as the waist to hip circumference.
  Overnight fasting blood samples were collected in tubes containing liquid EDTA; the samples were centrifuged at -4°C and maintained at -80°C until assayed. FBG was assayed using the glucose oxidase method. UA, TC, TG, LDL-C and HDL-C concentrations were determined enzymatically.

CONTACTS AND LOCATIONS:
Overall Officials: Deng Wuquan, PHD, Study Director — Southwest Hospital, China

REFERENCES:
- [Derived] Deng W, Li C, Zhang Y, Zhao J, Yang M, Tian M, Li L, Zheng Y, Chen B, Yang G. Serum C1q/TNF-related protein-3 (CTRP3) levels are decreased in obesity and hypertension and are negatively correlated with parameters of insulin resistance. Diabetol Metab Syndr. 2015 Apr 10;7:33. doi: 10.1186/s13098-015-0029-0. eCollection 2015. PMID 25878729
- See also: Implication of Progranulin and C1q/TNF-Related Protein-3 (CTRP3) on Inflammation and Atherosclerosis in Subjects with or without Metabolic Syndrome — http://www.plosone.org/article/info%3Adoi%2F10.1371%2Fjournal.pone.0055744
- See also: Identification of Adipokine Clusters Related to Parameters of Fat Mass, Insulin Sensitivity and Inflammation — http://www.plosone.org/article/info%3Adoi%2F10.1371%2Fjournal.pone.0099785